CLINICAL TRIAL: NCT06622265
Title: Multi-phase, Prospective, Multicenter, Non-interventional, Pre-market, Non-randomized, Open-label Study to Evaluate the Clinical Performance of the WHOOP ECG Feature
Brief Title: WHOOP ECG Software Performance Assessment Study
Status: Completed | Type: Observational
Sponsor: Whoop Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECG1-008
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Subjects whose ECG is interpreted as normal sinus rhythm during the screening assessment
  Interventions: Device: Electrocardiogram recording
- Cohort 2: Subjects whose ECG is interpreted as atrial fibrillation during the screening assessment
  Interventions: Device: Electrocardiogram recording

INTERVENTIONS:
Device: Electrocardiogram recording — ECG recording with investigational device

SUMMARY:
The purpose of the study is to evaluate the performance of ECG classification algorithms and their ability to classify heart rhythms into multiple categories of rhythms and heart rates.

DETAILED DESCRIPTION:
Atrial fibrillation (Afib) is the most common cardiac arrhythmia in the United States, affecting up to one in four individuals across the lifespan, and is associated with substantial morbidity and mortality. Fifteen percent of strokes in the United States are attributable to Afib, and nearly 20% of these occur in individuals with no prior Afib history. Because Afib is often paroxysmal, one-time screening is unlikely to capture those at risk. Thus, there has been an increasing interest in leveraging monitoring for Afib via wearable devices, which provide a novel method to monitor Afib and determine the burden of Afib in the general population.

The primary objective of this study is to assess the sensitivity and specificity of the investigation device (WHOOP ECG Feature) for the detection of Afib as compared to a gold-standard reference (12-Lead ECG Holter Device).

ELIGIBILITY:
Inclusion Criteria:

* Aged 22 years or older.
* Ability to provide informed consent.
* Willing to participate and to follow the procedures per the Principal Investigator's instructions.
* Resided in the United States.
* Wrist circumference: 130 mm to 245 mm at band wear position.
* Previous medical history of persistent, paroxysmal, or permanent or chronic AF and being in AF at time of enrollment (AF cohort only).
* No known history of AF and being in normal sinus rhythm at the time of enrollment (NSR cohort only).

Exclusion Criteria:

-Subjects with an implantable pacemaker device or implantable cardioverter- defibrillator device.

* Medical history of a life-threatening cardiac arrhythmia, e.g., ventricular tachycardia or fibrillation.
* Any known allergies to medical adhesives, isopropyl alcohol, or ECG patch.
* Any known allergy or sensitivity to thermoplastics, metals with physical vapor deposition (PVD) coatings or Elastane used in the wrist fitness devices.
* Clinically significant body tremors that compromise study measurements.
* Pregnant at the time of enrollment.
* Any physical disability that prevents safe and adequate testing.
* Physical or medical impairments that preclude exercise testing, including, but not limited to, back pain and leg claudication.
* Mental impairment as determined by the Investigator, or designee.
* Subjects with any medical history, physical examination finding, vital sign or other finding or assessment that could compromise subject safety, study integrity or accurate assessment of study objectives. This includes, but is not limited to, known untreated medical conditions that may be considered clinically significant, such as significant anemia, electrolyte imbalance, untreated or uncontrolled thyroid disease, and open wound(s) in the area of test band positioning.
* Vital sign measurements, medical history or physical examination finding that makes the subject inappropriate for participation according to the Investigator.
* Scarring, tattoos, large, pigmented moles, or other skin pathology in the area of sensor location.
* Severe skin conditions on either wrist, that would preclude wearing the sensor. Severe symptomatic skin injury, disorder, allergy, or disease such as eczema, rosacea, impetigo, dermatomyositis or contact dermatitis on wrist or other areas where sensors or electrodes would be placed.
* Clinically significant hand tremors as judged by the Investigator.
* Participated in phase 1 of the study (Only for phase 2 cohort).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adults seen in primary care and cardiology clinics associated with a single health system or subjects recruited through study advertisement. The prospective cohort will comprise two distinct populations - individuals with a known history of persistent atrial fibrillation and individuals without a history of cardiac arrhythmia of any kind.
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Specificity of the WHOOP ECG Feature for detection of sinus rhythm | 1 Day
  Specificity is defined as the True Negatives/(True Negatives + False Positives). A true normal sinus rhythm reading will have a 12-lead ECG reading consistent with normal sinus rhythm. A true negative is defined as individuals who have normal sinus rhythm reported on their ECGs from both the WHOOP ECG Feature and the 12-lead ECG Holter Device. A false positive is defined as individuals who receive an ECG with atrial fibrillation by the WHOOP ECG Feature but their 12-lead ECG has an atrial fibrillation determined by adjudication.
Sensitivity of the WHOOP ECG Feature for detection of atrial fibrillation | 1 Day
  Sensitivity is defined as the True Positives/(True Positives + False Negatives). A true atrial fibrillation reading will have an 12-lead ECG reading consistent with atrial fibrillation. A true positive is defined as individuals who have atrial fibrillation reported on their WHOOP ECGs and on the 12-lead ECG from the Holter Device. A false negative is defined as individuals who receive an ECG with atrial fibrillation with the 12-lead ECG as determined by adjudication but their WHOOP ECG Feature determination is Normal Sinus Rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Early, M.D., Principal Investigator — Iqvia Pty Ltd
Locations (7):
- United States (7):
  - HOPE Research Institute, Phoenix, Arizona
  - Valley Clinical Trials, Covina, California
  - Valley Clinical Trials, Northridge, California
  - Flourish Research, Winter Park, Florida
  - IQVIA, Lenexa, Kansas
  - Fairview Frontiers, Saint Paul, Minnesota
  - Eximia Research-NC, LLC, Raleigh, North Carolina